CLINICAL TRIAL: NCT00129545
Title: WATCHMAN Left Atrial Appendage System for Embolic PROTECTion in Patients With Atrial Fibrillation (PROTECT AF)
Brief Title: WATCHMAN Left Atrial Appendage System for Embolic PROTECTion in Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ST1021 and ST1055
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; AF; A Fib; Stroke; Coumadin; Warfarin; Blood thinning medication; transient ischemic attack (TIA); WATCHMAN; Left atrial appendage; LAA isolation; LAA occlusion
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Attack, Transient | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WATCHMAN (Experimental): Implant of WATCHMAN Left Atrial Appendage Closure Technology
  Interventions: Device: WATCHMAN Left Atrial Appendage Closure Technology
- Warfarin control (Active Comparator): Subjects are treated with current standard of care Oral Anticoagulation Therapy with Warfarin
  Interventions: Drug: Warfarin
- Roll-in (Other): Implant of WATCHMAN Left Atrial Appendage Closure Technology. Up to 3 non-randomized subjects per site, these subjects were not included in the primary analysis.
  Interventions: Device: WATCHMAN Left Atrial Appendage Closure Technology

INTERVENTIONS:
Device: WATCHMAN Left Atrial Appendage Closure Technology — Implant of WATCHMAN Left Atrial Appendage Closure Technology
  Other Names: WATCHMAN
  Arms: Roll-in; WATCHMAN
Drug: Warfarin — Subjects receive warfarin
  Other Names: Coumadin
  Arms: Warfarin control

SUMMARY:
This is a multi-center, prospective, randomized study, stratified by center, comparing the WATCHMAN device to long term warfarin therapy, demonstrating that the treatment arm is non-inferior to the control arm. This study was amended to allow for a non-randomized arm and increased enrollment.

DETAILED DESCRIPTION:
The WATCHMAN device is designed to be permanently implanted distal to the ostium of the left atrial appendage (LAA) to trap potential emboli before they exit the LAA.

ELIGIBILITY:
Inclusion Criteria:

* Patient has paroxysmal, persistent or permanent non-valvular atrial fibrillation (AF)
* Eligible for long term warfarin
* CHADS score >= 1 [congestive heart failure (CHF), history of high blood pressure, 75 years of age or older, diabetes, prior stroke or transient ischemic attack (TIA)]

Exclusion Criteria:

* Contraindicated for warfarin
* Contraindicated for aspirin or clopidogrel (Plavix)
* Congestive heart failure (CHF) Class 4
* Implanted mechanical valve
* Atrial septal or Patent Foramen Ovale (PFO) device
* Platelets < 100,000 or hemoglobin < 10
* Left ventricular ejection fraction (LVEF) < 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2005-02; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Holmes, MD, Principal Investigator — Mayo Clinic
Locations (62):
- United States (58):
  - Advanced Cardiac Specialists, Gilbert, Arizona
  - Arizona Arrhythmia, Scottsdale, Arizona
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - Los Angeles Cardiology Associates, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Orange County Heart, Orange County, California
  - UC Davis Medical Center, Sacramento, California
  - St. John's Hospital / Pacific Heart, Santa Monica, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Bay Heart Group, Tampa, Florida
  - Emory University Midtown Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - North Shore University, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Prairie Education Research Cooperative, Springfield, Illinois
  - Baptist Hospital West, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - William Beaumont, Royal Oak, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - University of Mississippi Healthcare Center, Jackson, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New York University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Summa Health System, Akron, Ohio
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Harrisburg Hospital / Associated Cardiology, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - Moffitt Heart & Vascular, Wormleysburg, Pennsylvania
  - Mercy Medical Center West, Knoxville, Tennessee
  - St. Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - St. Lukes Episcopal Hospital, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Na Homolce, Prague, Czechia
- Germany (3):
  - Krankenhaus der Barmherzige Bruder, Regensburg, Bavaria
  - Cardiovasculares Centrum Frankfurt - Sankt Katharinen, Frankfurt am Main, Hesse
  - Herzzentrum, Leipzig

REFERENCES:
- [Derived] Dukkipati SR, Holmes DR Jr, Doshi SK, Kar S, Singh SM, Gibson D, Price MJ, Natale A, Mansour M, Sievert H, Houle VM, Allocco DJ, Reddy VY. Impact of Peridevice Leak on 5-Year Outcomes After Left Atrial Appendage Closure. J Am Coll Cardiol. 2022 Aug 2;80(5):469-483. doi: 10.1016/j.jacc.2022.04.062. PMID 35902169
- [Derived] Brouwer TF, Whang W, Kuroki K, Halperin JL, Reddy VY. Net Clinical Benefit of Left Atrial Appendage Closure Versus Warfarin in Patients With Atrial Fibrillation: A Pooled Analysis of the Randomized PROTECT-AF and PREVAIL Studies. J Am Heart Assoc. 2019 Dec 3;8(23):e013525. doi: 10.1161/JAHA.119.013525. Epub 2019 Nov 22. PMID 31752643
- [Derived] Price MJ, Reddy VY, Valderrabano M, Halperin JL, Gibson DN, Gordon N, Huber KC, Holmes DR Jr. Bleeding Outcomes After Left Atrial Appendage Closure Compared With Long-Term Warfarin: A Pooled, Patient-Level Analysis of the WATCHMAN Randomized Trial Experience. JACC Cardiovasc Interv. 2015 Dec 28;8(15):1925-1932. doi: 10.1016/j.jcin.2015.08.035. Epub 2015 Nov 25. PMID 26627989
- [Derived] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Derived] Alli O, Doshi S, Kar S, Reddy V, Sievert H, Mullin C, Swarup V, Whisenant B, Holmes D Jr. Quality of life assessment in the randomized PROTECT AF (Percutaneous Closure of the Left Atrial Appendage Versus Warfarin Therapy for Prevention of Stroke in Patients With Atrial Fibrillation) trial of patients at risk for stroke with nonvalvular atrial fibrillation. J Am Coll Cardiol. 2013 Apr 30;61(17):1790-8. doi: 10.1016/j.jacc.2013.01.061. Epub 2013 Feb 28. PMID 23500276
- [Derived] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Derived] Reddy VY, Holmes D, Doshi SK, Neuzil P, Kar S. Safety of percutaneous left atrial appendage closure: results from the Watchman Left Atrial Appendage System for Embolic Protection in Patients with AF (PROTECT AF) clinical trial and the Continued Access Registry. Circulation. 2011 Feb 1;123(4):417-24. doi: 10.1161/CIRCULATIONAHA.110.976449. Epub 2011 Jan 17. PMID 21242484
- [Derived] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- See also: Sponsor website — http://www.atritech.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Roll-in: Investigational centers were allowed up to 3 roll in subjects before initiating the randomization phase
- WATCHMAN: Randomized to receive implantation of the WATCHMAN left atrial appendage (LAA) closure Technology
- WARFARIN: Randomized to receive Warfarin control
Period: Overall Study
Arm/Group | Roll-in | WATCHMAN | WARFARIN
Started | 93 | 463 (2:1 randomization WATCHMAN to warfarin) | 244
Completed | 67 | 299 | 133
Not Completed | 26 | 164 | 111
Not completed — Death | 5 | 60 | 44
Not completed — Withdrawal by Subject | 3 | 18 | 44
Not completed — Lost to Follow-up | 2 | 22 | 13
Not completed — Physician Decision | 0 | 3 | 10
Not completed — Device not implanted | 16 | 61 | 0

BASELINE CHARACTERISTICS:
Population: 2:1 randomazation, outcome analysis excludes the 93 subjects in the Roll-in arm
Groups:
- WATCHMAN: WATCHMAN Left Atrial Appendage Closure Technology:
- Warfarin Control: Subjects were treated with current standard of care Oral Anticoagulation Therapy with Warfarin
- Roll-in: Subjects received WATCHMAN Left Atrial Appendage Closure Technology but were not included in the outcome analysis
- Total: Total of all reporting groups
Arm/Group | WATCHMAN | Warfarin Control | Roll-in | Total
Number analyzed (Participants) | 463 | 244 | 93 | 800
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.8) | 72.7 (9.2) | 72.2 (8.9) | 72.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 73 | 28 | 238
  Male | 326 | 171 | 65 | 562
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4 | 1 | 0 | 5
  Black/African American | 6 | 5 | 3 | 14
  Caucasian | 425 | 222 | 87 | 734
  Hispanic/Latino | 25 | 15 | 3 | 43
  Hawaiian/Pacific Islander | 1 | 1 | 0 | 2
  other | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 382 | 201 | 87 | 670
  Czech Republic | 19 | 10 | 3 | 32
  Germany | 62 | 33 | 3 | 98

OUTCOME MEASURES:

1. Primary Outcome: Composite of Stroke, Systemic Embolism and Cardiovascular or Unexplained Death
Description: A Bayesian model allowed for sequential evaluation of the primary endpoints, event rates reported per 100 patient-years (calculated as 100*N events/Total patient-years)
Time Frame: 5 years
Population: event rates reported per 100 patient-years (calculated as 100*N events/Total patient-years) total patient years 2717, 95% Credible Intervals per predefined Bayesian Statistics
  Roll-in subjects were not included in the primary outcome analysis per study design.
Measure: Number (95% Confidence Interval); unit: events per 100 pt yrs
Groups:
- Implantable Device: Implantable WATCHMAN Left ATrial Appendage Occlusion Device
  WATCHMAN Left Atrial Appendage Closure Technology: Implant of WATCHMAN Left Atrial Appendage Closure Technology
Arm/Group | Implantable Device | Warfarin Control
Number analyzed (Participants) | 463 | 244
events per 100 pt yrs | 2.2 [1.7 to 3.1] | 3.7 [2.4 to 4.8]
Statistical Analysis 1: Comparison: Implantable Device vs Warfarin Control; Test type: Non-Inferiority or Equivalence — The posterior probability of non-inferiority is defined as the probability that the event rate for the Device group is less than twice that for the Control group. This probability was required to be greater than 0.975 for a finding of non-inferiority. The criterion for non-inferiority was consistently met at each analysis time point demonstrating the Device group is non-inferior to the Control group; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.42 to 1.07] — Relative Risk calculated as Device Rate over Control rate, with 95% Credible Intervals

2. Primary Outcome: The Occurrence of Life-threatening Events, Including Device Embolization or Serious Bleeding Events
Description: Serious bleeding events evaluated by the Clinical Events Committee included pericardial effusion requiring drainage, cranial bleeding events due to any source, gastrointestinal bleeds requiring transfusion, and any bleeding related to the device or procedure that necessitates an operation.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 pt-yrs
Arm/Group | Implantable Device | Warfarin Control
Number analyzed (Participants) | 463 | 244
Events per 100 pt-yrs | 3.5 [2.7 to 4.5] | 3.2 [2.1 to 4.4]

3. Secondary Outcome: Procedure Success
Description: Implant procedure success is defined as the delivery and release of a WATCHMAN Device into the LAA.
Time Frame: Initial implant procedure
Population: 14 subjects did not have an implant procedure attempted
Measure: Number; unit: percentage of implant attempts
Groups:
- WATCHMAN: Implantable WATCHMAN Left ATrial Appendage Occlusion Device
  Implant of WATCHMAN Left Atrial Appendage Closure Technology
Arm/Group | WATCHMAN
Number analyzed (Participants) | 449
percentage of implant attempts | 90.9

ADVERSE EVENTS:
Time Frame: 5 years
Description: electronic case report form (e-CRF) completion by sites, followed by independent Clinical Events Committee (CEC) adjudication
Groups:
- WATCHMAN: Randomized to receive implantation of the WATCHMAN LAA closure Device
Arm/Group | Roll-in | WATCHMAN | WARFARIN
Serious Adverse Events (participants affected / at risk) | 29/93 | 143/463 | 70/244
Other Adverse Events (participants affected / at risk) | 19/93 | 71/463 | 17/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-in (N=93) | WATCHMAN (N=463) | WARFARIN (N=244)
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (4)
Arrhythmias (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
AV Fistula (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Bleeding from Varicose Veins (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising - Hematoma (Vascular disorders) | 2 (2) | 5 (5) | 0 (0)
Cardiac Perforation (Cardiac disorders) | 1 (1) | 7 (7) | 0 (0)
Cranial Bleed (Vascular disorders) | 1 (1) | 4 (4) | 1 (1)
Death (General disorders) | 5 (5) | 59 (59) | 44 (44)
Device Embolization (Investigations) | 0 (0) | 3 (4) | 0 (0)
Device Thrombus (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 9 (12) | 26 (32) | 22 (27)
Hematuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Major Bleed Requiring Transfusion (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Oral Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Other Study Related (Investigations) | 4 (4) | 17 (18) | 2 (2)
Pericardial Effusion with Cardiac Tamponade (Cardiac disorders) | 4 (4) | 13 (13) | 0 (0)
Pericardial Effusion-Serious (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Stroke - Hemorrhagic (Nervous system disorders) | 0 (0) | 3 (3) | 10 (10)
Stroke - Ischemic (Nervous system disorders) | 5 (5) | 24 (26) | 10 (11)
Systemic Embolization (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1) | 5 (5) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roll-in (N=93) | WATCHMAN (N=463) | WARFARIN (N=244)
Air Embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Allergic Reaction to Contrast Media (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
AV Fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Bleeding from Varicose Veins (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising - Hematoma (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
Device Thrombus (Investigations) | 2 (2) | 14 (15) | 0 (0)
Epistaxis (Vascular disorders) | 4 (4) | 11 (13) | 5 (5)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Inability to Move or Retrieve Device (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Other Non-Study Related (General disorders) | 0 (0) | 2 (2) | 0 (0)
Other Study Related (Investigations) | 9 (9) | 19 (20) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 3 (3) | 10 (10) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 3 (5) | 5 (5)
Stroke - Ischemic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Vasovagal Reactions (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less